CLINICAL TRIAL: NCT06543342
Title: Bystander Intervention for Hazardous Drinking
Acronym: DISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Nancy Barnett, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AA025456
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Hazardous Behavior; Alcohol Consequences
MeSH Terms: conditions — Dangerous Behavior

STUDY DESIGN:
Intervention Model Description: 2-group trial in which one group serves as intervention recipients and one as assessment-only controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bystander Brief Motivational Intervention (Experimental): Two 2-hour in person sessions focusing on identifying alcohol risks among peers, determining optimal bystander strategies to use, and identifying personal barriers to intervening.
  Interventions: Behavioral: Bystander Brief Motivational Intervention
- Assessment Control (No Intervention): Comparison group selected using the same criteria but receive no intervention.

INTERVENTIONS:
Behavioral: Bystander Brief Motivational Intervention — Group-based interactive intervention, conducted in two sessions, including multiple tasks and exercises to identify different levels of risk behavior, different types of strategies, and practicing responding to different scenarios. Personal goals for helping friends stay safe, and identifying whether intervention as a bystander was successful are included.
  Arms: Bystander Brief Motivational Intervention

SUMMARY:
The objective of this treatment development grant is to create an innovative and efficacious alcohol intervention for emerging adults using features from three theoretically sound and empirically supported approaches. A set of students will be engaged to serve as peer leaders to assist in reducing hazardous drinking behavior among their peers. This new intervention, a Bystander Brief Motivational Intervention (BBMI) spans Stages 1A and 1B of the stage model of behavioral therapies research and will utilize qualitative methods, an open trial, and a small controlled pilot trial within the targeted college community.

DETAILED DESCRIPTION:
The objective of this treatment development grant is to create an innovative and efficacious alcohol intervention for emerging adults using features from three theoretically sound and empirically supported approaches. Established elements from Bystander Intervention (awareness of the problem, addressing pluralistic ignorance, skill building), Brief Motivational Intervention (client-centered foundation, corrective information about community norms, protective behavioral strategies) and Social Network Analysis (measuring network ties, identifying the influence of network members), will be integrated into a brief intervention that pays particular attention to the connectedness of residents in dormitory social networks. Social network analytic methods will be used to assess the primary peer network (the college residence) and a set of individuals exposed to others drinking risks will be identified to receive the intervention. This set of students will be engaged to serve as peer leaders to assist in reducing hazardous drinking behavior among their peers. This new intervention, a Bystander Brief Motivational Intervention (BBMI) spans Stages 1A and 1B of the stage model of behavioral therapies research and will utilize qualitative methods, an open trial, and a small controlled pilot trial within the targeted college community.

ELIGIBILITY:
Inclusion Criteria:

* First-year students in one of two residence halls. The subset of participants who were selected for intervention or control had to have been exposed to others who showed risk signs in the past month.

Exclusion Criteria:

* None

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Exposure to the Hazardous Drinking of Others | 1 month and 3 months
  Number of risk signs observed in peers -validated measure
The Bystanders to Alcohol Risk Scale - Strategies | 1 month and 3 months
  Number of strategies used to help others - validated measure
Alcohol Bystander Readiness to Help | 1 month and 3 months
  Self-perception of readiness to help others in different situations - measure validation underway

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No